CLINICAL TRIAL: NCT01248546
Title: Digital Breast Tomosynthesis in the Oslo Mammography Screening Program
Brief Title: Tomosynthesis in the Oslo Breast Cancer Screening Program
Acronym: DBT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Institute of Public Health (Other Government); Hologic, Inc. (Industry)
Responsible Party: Principal Investigator, Per Skaane, professor dr. med., Oslo University Hospital
Other Study IDs: 2010/144 (REK)
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Recall Rate; Cancer Detection Rate; False Positive Rate; Positive Predictive Value
Keywords: Breast cancer; Computer-aided detection; Mammography screening; Digital breast tomosynthesis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Digital mammography
  Interventions: Procedure: Digital breast tomosynthesis

INTERVENTIONS:
Procedure: Digital breast tomosynthesis — The participants included in the trial will have an additional radiation exposure for breast tomosynthesis

SUMMARY:
The Digital Breast Tomosynthesis (DBT) in the Oslo Mammography Screening Program will include women aged 50 to 69 years invited to the population-based mammography-screening program. All women attending the screening unit will be asked if they want to attend the trial. If so, they will be informed about the project, the technique, and the additional compression and radiation dose. All mammographic examinations of women attending the trial will be independently interpreted by four radiologists. Since the trial is part of the official Norwegian Breast Cancer Screening Program (NBCSP), the interpretations will be carried out on-line into the national screening database of the NBCSP. The study will include independent reading of conventional digital (2D) mammograms, 2D plus computer-aided detection (CAD), 2D plus DBT, and synthetic 2D plus DBT. There will be a common consensus meeting for all examinations having a positive score. Recalls and diagnostic work-up will be according to daily practice at the Oslo University Hospital Ullevaal and the guidelines of the NBCSP.

Outcome measures will use performance indicators for organized screening programs, including recall rate, false positive scores, cancer detection rate, positive predictive values, and cancer characteristics for the individual readers of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Women 50 to 69 years who have signed the informed consent

Exclusion Criteria:

* Women with pacemaker, implants, and severely disabled

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women aged 50 to 69 years attending the national breast cancer screening program who sign an informed consent regarding participation in the trial
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Screening performance indicators | From Nov. 22, 2010 to Dec. 31, 2012

SECONDARY OUTCOMES:
Interval cancer rate | From Nov. 23, 2010 to Dec. 31, 2014

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Ulleval, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Skaane P, Sebuodegard S, Bandos AI, Gur D, Osteras BH, Gullien R, Hofvind S. Performance of breast cancer screening using digital breast tomosynthesis: results from the prospective population-based Oslo Tomosynthesis Screening Trial. Breast Cancer Res Treat. 2018 Jun;169(3):489-496. doi: 10.1007/s10549-018-4705-2. Epub 2018 Feb 10. PMID 29429017
- [Derived] Skaane P, Bandos AI, Gullien R, Eben EB, Ekseth U, Haakenaasen U, Izadi M, Jebsen IN, Jahr G, Krager M, Niklason LT, Hofvind S, Gur D. Comparison of digital mammography alone and digital mammography plus tomosynthesis in a population-based screening program. Radiology. 2013 Apr;267(1):47-56. doi: 10.1148/radiol.12121373. Epub 2013 Jan 7. PMID 23297332